CLINICAL TRIAL: NCT02282137
Title: 68Ga-PSMA (ProstaMedix™) PET-CT Scan for Diagnosis and Management of Prostate Cancer
Brief Title: 68Ga-PSMA PET-CT Scan for Diagnosis and Management of Prostate Cancer
Acronym: PSMA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ebrahim Delpassand (Other)
Collaborators: Radiomedix, Inc. (Industry); Excel Diagnostics and Nuclear Oncology Center (Other)
Responsible Party: Sponsor-Investigator, Ebrahim Delpassand, Chairman and Medical Director, Radio Isotope Therapy of America
Organization: Radio Isotope Therapy of America (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Ga PSMA124388; IND124388 (Other: US Food and Drug Administration)
Record Dates: First submitted 2014-10-27; First posted 2014-11-04 (Estimated); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; PET / CT; Ga-PSMA
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 68Ga-PSMA (Experimental): Evaluation of concordance and discordance between the results of 68Ga-PSMA PET/CT and other available conventional imaging modalities (such as CT, MRI, FDG, NaF scan), histology or follow up.
  Interventions: Drug: 68Ga-PSMA

INTERVENTIONS:
Drug: 68Ga-PSMA — Patients with suspected prostate cancer recurrence and non-informative bone scintigraphy, computerized tomography (CT) or magnetic resonance imaging (MRI). Suspected prostate recurrence is based upon elevated blood prostate specific antigen (PSA) levels following initial therapy.
  Other Names: 68Ga-HBED-CC-PSMA

SUMMARY:
This is a phase II clinical trial study to show how well the 68Ga-PSMA-11 (ProstaMedix™) PET-CT scan works in detecting tumor location and size in patients with suspected or confirmed prostate cancer, as well as prostate cancer that may have come back in patients with elevated PSA ( a prostate-specific antigen tumor marker) after initial treatment.

DETAILED DESCRIPTION:
68Ga-PSMA-11 is a radioactive imaging contrast agent for use in PET CT scan that seeks to identify prostate cancer cells that have a specific protein target called prostate-specific membrane antigen (PSMA) on their surface. PET and CT make computerizing pictures of areas inside the body where the radioactive substance is lighting up. 68Ga-PSMA-11 PET / CT may be able to see smaller tumors than standard imaging and may help determine whether prostate cancer has come back and where it is in the body.

A 68Ga-PSMA-11 PET / CT scan may help doctors to better detect the location, extent, and characteristics of the tumor, allowing improved planning of subsequent therapy

ELIGIBILITY:
Inclusion Criteria

General requirements:

1. Karnofsky performance status of ≥50 (or ECOG/WHO equivalent).
2. Age > 18 years .
3. Ability to understand a written informed consent document, and the willingness to sign it.
4. i. inclusion criteria specific for the pre-prostatectomy group:

   * Biopsy proven prostate adenocarcinoma.
   * Planned prostatectomy with lymph node dissection.
   * Intermediate to high-risk disease (as determined by elevated PSA [PSA>10], T-stage [T2b or greater], Gleason score [Gleason score > 6] or other risk factors).

4. ii. inclusion criteria specific for biochemical recurrence group:

* Histopathological proven prostate adenocarcinoma.
* Rising PSA after definitive therapy with prostatectomy or radiation therapy (external beam or brachytherapy).

  1. Post radical prostatectomy (RP) - AUA recommendation, PSA greater than or equal to 0.2 ng/mL measured more than 6 weeks after RP.
  2. Post-radiation therapy -ASTRO-Phoenix consensus definition, Nadir + greater than or equal to 2 ng/mL rise in PSA 5. Diagnostic CT or MRI as part of the PET study or performed within one month of PSMA PET

Exclusion Criteria

General requirements:

1. Patients not capable of getting PET study due to weight, claustrophobia, or inability to lay still for the duration of the exam.
2. Contraindication to furosemide administration including prior allergy or adverse reaction to furosemide or sulfa drugs. (Note: This exclusion criterion can be removed if Furosemide is omitted as part of the PET imaging protocol if a second-generation scatter correction is available for the used PET device).
3. i. Exclusion criteria specific for the pre-prostatectomy group: Neoadjuvant chemotherapy or radiation therapy prior to prostatectomy, including focal ablation techniques (HiFu) within the last 2 months.

3. ii. Exclusion criteria specific for biochemical recurrence group:

* Investigational therapy for prostate cancer for less than 2 months.
* Prior history of any other malignancy within the last 2 years, other than skin basal cell or cutaneous superficial squamous cell carcinoma that has not metastasized and superficial bladder cancer.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2015-05 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The sensitivity of 68Ga-PSMA-11 PET for detection of tumor location. | 12 months
  The sensitivity of 68Ga-PSMA-11 PET to detect tumor location and metastases in patients with biopsy confirmed diagnosis.tumor location confirmed by histopathology/biopsy and conventional imaging follow-up.

SECONDARY OUTCOMES:
Detection rates of 68Ga-PSMA-11 PET in patients with different PSA value | 12 months
  Detection rates of 68Ga-PSMA-11 PET in patients with different PSA value (0.2 - <0.5, 0.5 - <1.0, 1.0 - <2.0, 2.0 - <5.0, 5.0).

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo Nunez, MD, Principal Investigator — Excel Diagnostics and Nuclear Oncology Center
Locations (1):
- Radio- Isotope Therapy of America, Houston, Texas, United States